CLINICAL TRIAL: NCT03605849
Title: An Open-label, 52-Week, Multicenter Trial Evaluating the Long-term Safety and Tolerability of Centanafadine Sustained-Release Tablets in Adults With Attention-Deficit/Hyperactivity Disorder
Brief Title: A Trial Evaluating the Long-term Safety and Tolerability of Centanafadine Sustained-release Tablets in Adults With Attention-Deficit/Hyperactivity Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 405-201-00015
Record Dates: First submitted 2018-06-28; First posted 2018-07-30 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Attention Deficit Disorder; Attention Deficit Hyperactivity Disorder
Keywords: Centanafadine; ADD; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 1-(naphthalen-2-yl)-3-azabicyclo(3.1.0)hexane

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Centanafadine (Experimental): 400 mg total daily dose
  Interventions: Drug: Centanafadine SR

INTERVENTIONS:
Drug: Centanafadine SR — 200mg, BID, oral tablets
  Other Names: EB-1020

SUMMARY:
This study evaluated the long-term safety and tolerability of centanafadine sustained-release (SR) tablets, administered twice daily (BID) in the treatment of adults with attention deficit hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
This open-label study assessed the overall safety and tolerability of 400 mg total daily dose centanafadine SR tablets in participants, over the course of approximately 52 weeks. This study has accepted rollover participants from both the 405-201-00013 and 405-201-00014 trials. For individuals that did not participate in one of the studies mentioned above, they will be able to enroll if they meet the inclusion criteria as outlined below.

ELIGIBILITY:
De Novo Participants [De Novo Enrollment has ended 20Sep2019].

Inclusion Criteria:

* De novo participants must meet the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for ADHD (including predominantly inattentive presentation, hyperactive presentation, or combined presentation) as confirmed by the Adult ADHD Clinical Diagnostic Scale (ACDS) Version 1.2. To confirm that ADHD is the primary diagnosis, the Mini International Neuropsychiatric Interview (MINI) will be used to identify and exclude other psychiatric conditions which would preclude enrollment.
* Participants are 18 to 55 years of age, inclusive, at the time of consent.
* Participants have BMI of 18 to 40, inclusive
* Participants are willing to discontinue all prohibited psychotropic medications starting from the time of signing the informed consent and up to the 10-day safety follow-up period.

Exclusion Criteria:

* Participants has a DSM-5 diagnosis of Other Specified or Unspecified Attention-Deficit/Hyperactivity Disorder as confirmed by ACDS Version 1.2.
* Participant has a current comorbid psychiatric disorder that is either controlled with medications prohibited in this trial or is uncontrolled and associated with significant symptoms, including but not limited to: a current major depressive episode (per DSM-5 criteria), current symptoms (past 90 days) meeting the DSM-5 criteria for a diagnosis of generalized anxiety disorder, obsessive compulsive disorder, panic disorder, or posttraumatic stress disorder, as established by the MINI. NOTE: Participants with mild mood or anxiety symptoms that do not meet criteria for diagnosis, who do not require treatment based on the Investigator's assessment, and do not confound efficacy or safety assessments in the opinion of the examining Investigator, may be included.
* Participants that have a positive alcohol test (via breathalyzer or blood), a positive drug screen for cocaine, or other illicit drugs (excluding marijuana). Participants with a positive drug screen for confirmed prescription medications at baseline will not be permitted to continue participation in Trial 405-201-00015. NOTE: Participants that tested positive for marijuana may be permitted to be enrolled if they have no evidence of a substance use disorder, and if they agree to refrain from use for the duration of the trial. Allowance for participants testing positive for marijuana at screening require explicit approval from the medical monitor.

Rollover Participants: Rollover Enrollment has ended 28Aug2020.

Inclusion Criteria:

* Participants who completed the double-blind treatment period and 7-day follow-up after last dose of investigational medicinal product (IMP) in double-blind trials and who, in the opinion of the investigator, could potentially benefit from centanafadine for ADHD.

Exclusion Criteria:

* Participants who, during the double-blind phase 3 trial experienced, in the opinion of the investigator, poor tolerability to trial medication or whose safety assessments resulted in new concerns that would suggest the participant may not be appropriate for a 52-week treatment with trial medication.
* Participants who have re-initiated any therapy for adult ADHD during the 7-day follow-up period after the final treatment visit of the double-blind phase 3 trial.
* Participants that have a positive alcohol test (via breathalyzer or blood), a positive drug screen for cocaine, or other illicit drugs (excluding marijuana). Participants with a positive drug screen for confirmed prescription medications at baseline will not be permitted to continue participation in Trial 405-201-00015. NOTE: Participants that test positive for marijuana may not be permitted to rollover into the open label study, and must agree to refrain from use for the duration of the open label trial. Allowance for participants testing positive for marijuana at time of rollover requires explicit approval from the medical monitor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 662 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding sites, contact 844-687-8522, Culver City, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com
URL: http://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in the United States from 14 February 2019 to 07 September 2021. A total of 662 participants were enrolled in the study. Out of 662 participants, 653 participants received the study treatment.
Pre-assignment Details: A total of 662 participants were treated in this study, 494 participants from parent studies (405-201-00013 and 405-201-00014) &168 new participants joined in this current study. As pre-specified in Statistical analysis plan (SAP) data was analyzed by the parent studies (405-201-00013 and 405-201-00014) treatment groups for rollover participants and centanafadine SR 400mg for denovo participants. Data from the 2 parent studies was analyzed and reported in combined way for rollover participants.
Groups:
- Prior Centanafadine SR 200 mg: Participants who received centanafadine sustained release (SR) 200 milligrams (mg) in the parent double-blind phase 3 studies 405-201-00013 [NCT03605680] or 405-201-00014 [NCT03605836], received a total daily dose (TDD) of centanafadine SR 400 mg in current study, following a dose-escalation schedule. In the current study, participants received centanafadine SR tablets, orally, twice daily (BID) at a starting dose of 200 mg TDD on Day 1 through Day 7, followed by dose-escalation to 400 mg TDD from Day 8 up to Week 52.
- Prior Centanafadine SR 400 mg: Participants who received centanafadine SR 400 mg in the parent double-blind phase 3 studies 405-201-00013 [NCT03605680] or 405-201-00014 [NCT03605836], received centanafadine SR 400 mg TDD in current study, following a dose-escalation schedule. In the current study, participants received centanafadine SR tablets, orally, BID at a starting dose of 200 mg TDD on Day 1 through Day 7, followed by dose-escalation to 400 mg TDD from Day 8 up to Week 52.
- Prior Placebo: Participants who received placebo in the parent double-blind phase 3 studies 405-201-00013 [NCT03605680] or 405-201-00014 [NCT03605836], received centanafadine SR 400 mg TDD in current study, following a dose-escalation schedule. In the current study, participants received centanafadine SR tablets, orally, BID at a starting dose of 200 mg TDD on Day 1 through Day 7, followed by dose-escalation to 400 mg TDD from Day 8 up to Week 52.
- De Novo Centanafadine SR 400 mg: Participants who did not participate in the parent double-blind phase 3 studies 405-201-00013 [NCT03605680] or 405-201-00014 [NCT03605836], and who were eligible for this study received centanafadine SR 400 mg TDD in current study, following a dose-escalation schedule. In the current study, participants received centanafadine SR tablets, orally, BID at a starting dose of 200 mg TDD on Day 1 through Day 7, followed by dose-escalation to 400 mg TDD from Day 8 up to Week 52.
Period: Overall Study
Arm/Group | Prior Centanafadine SR 200 mg | Prior Centanafadine SR 400 mg | Prior Placebo | De Novo Centanafadine SR 400 mg
Started | 156 | 151 | 187 | 168
Safety Sample (Safety Sample comprised all participants who received at least 1 dose of investigational medicinal product (IMP).) | 154 | 149 | 184 | 166
Completed | 78 | 72 | 92 | 103
Not Completed | 78 | 79 | 95 | 65
Not completed — Adverse Event | 20 | 21 | 29 | 11
Not completed — Lack of Efficacy | 4 | 7 | 9 | 2
Not completed — Lost to Follow-up | 8 | 8 | 14 | 11
Not completed — Non-compliance With IMP | 6 | 5 | 2 | 1
Not completed — Protocol Deviation | 1 | 2 | 1 | 3
Not completed — Withdrawal by Subject | 33 | 28 | 30 | 28
Not completed — Site Terminated by Sponsor | 0 | 0 | 0 | 1
Not completed — Physician Decision | 2 | 1 | 2 | 1
Not completed — Enrolled, but not Treated | 2 | 2 | 3 | 2
Not completed — Other (COVID-19 Related) | 0 | 1 | 1 | 0
Not completed — Other (Not Related to COVID-19) | 2 | 4 | 4 | 5

BASELINE CHARACTERISTICS:
Population: Enrolled Sample comprised all participants who signed electronic informed consent form (ICF) for the trial.As prespecified in the SAP,data was analyzed based on the treatments(centanafadine SR 200mg, 400 mg or Placebo)received by the participants in the parent double-blind phase 3 trials(405-201-00013 or 405-201-00014),and the centanafadine SR 400 mg received by de novo participants during this study.Data from 2 parent studies was analyzed and reported in combined way for rollover participants.
Groups:
- Prior Centanafadine SR 200 mg: Participants who received centanafadine SR 200 mg in the parent double-blind phase 3 studies 405-201-00013 [NCT03605680] or 405-201-00014 [NCT03605836], received TDD of centanafadine SR 400 mg in current study, following a dose-escalation schedule. In the current study, participants received centanafadine SR tablets, orally, BID at a starting dose of 200 mg TDD on Day 1 through Day 7 , followed by dose-escalation to 400 mg TDD from Day 8 up to Week 52.
- Total: Total of all reporting groups
Arm/Group | Prior Centanafadine SR 200 mg | Prior Centanafadine SR 400 mg | Prior Placebo | De Novo Centanafadine SR 400 mg | Total
Number analyzed (Participants) | 156 | 151 | 187 | 168 | 662
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 156 | 151 | 187 | 168 | 662
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 76 | 76 | 94 | 92 | 338
  Male | 80 | 75 | 93 | 75 | 323
  Unknown | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 121 | 122 | 162 | 144 | 549
  Race: Black or African American | 19 | 21 | 16 | 10 | 66
  Race: American Indian or Alaska Native | 0 | 2 | 1 | 1 | 4
  Race: Asian | 7 | 1 | 6 | 9 | 23
  Race: Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Race: Other | 8 | 5 | 2 | 3 | 18
  Race: Unknown | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 34 | 36 | 35 | 50 | 155
  Ethnicity: Not Hispanic or Latino | 119 | 112 | 150 | 116 | 497
  Ethnicity: Other | 3 | 1 | 2 | 1 | 7
  Ethnicity: Unknown | 0 | 2 | 0 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 156 | 151 | 187 | 168 | 662

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Graded by Severity
Description: An AE is defined as any untoward medical occurrence in a patient or clinical trial participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. TEAEs are defined as AEs with an onset date on or after the first dose of IMP. They are all adverse events that started after the start of centanafadine; or if the event was continuous from baseline and was worsening, serious, study drug-related, or resulted in death, discontinuation, interruption or reduction of study therapy.
  TEAEs were graded on a 3-point scale and the intensity of an adverse experience was defined as follows: 1 = Mild: Discomfort noticed, but no disruption to daily activity, 2 = Moderate: Discomfort sufficient to reduce or affect normal daily activity, and 3 = Severe: Inability to work or perform normal daily activity.
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (Up to approximately Week 56)
Population: Safety Sample comprised all participants who received at least 1 dose of IMP. As prespecified in the SAP, data was analyzed based on the treatments (centanafadine SR 200mg, 400 mg or placebo) received by the participants in the parent double-blind phase 3 trials (405-201-00013 or 405-201-00014), and the centanafadine SR 400 mg received by de novo participants during this current study. Data from 2 parent studies was analyzed and reported in a combined way for rollover participants.
Measure: Count of Participants; unit: Participants
Groups:
- Prior Centanafadine SR 200 mg: Participants who received centanafadine SR 200 mg in the parent double-blind phase 3 studies 405-201-00013 [NCT03605680] or 405-201-00014 [NCT03605836], received centanafadine SR 400 mg TDD in current study, following a dose-escalation schedule. In current study, participants received centanafadine SR tablets, orally, BID at a starting dose of 200 mg TDD on Day 1 through Day 7, followed by dose-escalation to 400 mg TDD from Day 8 up to Week 52.
- Prior Centanafadine SR 400 mg: Participants who received centanafadine SR 400 mg in the parent double-blind phase 3 studies 405-201-00013 [NCT03605680] or 405-201-00014 [NCT03605836], received centanafadine SR 400 mg TDD in current study, following a dose-escalation schedule. In current study, participants received centanafadine SR tablets, orally, BID at a starting dose of 200 mg TDD on Day 1 through Day 7, followed by dose-escalation to 400 mg TDD from Day 8 up to Week 52.
- Prior Placebo: Participants who received placebo in the parent double-blind phase 3 studies 405-201-00013 [NCT03605680] or 405-201-00014 [NCT03605836], received centanafadine SR 400 mg TDD in current study, following a dose-escalation schedule. In current study, participants received centanafadine SR tablets, orally, BID at a starting dose of 200 mg TDD on Day 1 through Day 7, followed by dose-escalation to 400 mg TDD from Day 8 up to Week 52.
- De Novo Centanafadine SR 400 mg: Participants who did not participate in the parent double-blind phase 3 studies 405-201-00013 [NCT03605680] or 405-201-00014 [NCT03605836], and who were eligible for this study received centanafadine SR 400 mg TDD in current study, following a dose-escalation schedule. In current study, participants received centanafadine SR tablets, orally, BID at a starting dose of 200 mg TDD on Day 1 through Day 7, followed by dose-escalation to 400 mg TDD from Day 8 up to Week 52.
Arm/Group | Prior Centanafadine SR 200 mg | Prior Centanafadine SR 400 mg | Prior Placebo | De Novo Centanafadine SR 400 mg
Number analyzed (Participants) | 154 | 149 | 184 | 166
Participants
  Participants With TEAEs | 98 | 89 | 123 | 91
  Participants With Mild TEAE | 73 | 59 | 92 | 70
  Participants With Moderate TEAE | 58 | 53 | 75 | 50
  Participants With Severe TEAE | 2 | 4 | 7 | 3

2. Other Pre Specified Outcome: Adult ADHD Investigator Symptom Rating Scale (AISRS)
Description: 18-item scale with a total score range of 0 to 54 points. Composed of 2 subscales that can range from 0 to 27 points. A higher value represents a worse outcome. Efficacy endpoint. Results will be assessed to determine effectiveness of drug.
Time Frame: Up to 52 weeks or early termination
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Clinical Global Impression-Severity of Illness Scale (CGI-S)
Description: An observer-rated scale with a total score range of 0 to 7. A higher score represents a worse outcome.Efficacy endpoint. Results will be assessed to determine effectiveness of drug.
Time Frame: Up to 52 weeks or early termination
Reporting Status: Not Posted

4. Other Pre Specified Outcome: ADHD Impact Module - Adult (AIM-A)
Description: Scale composed of 3 subscales with a maximum score of 100. A lower score indicates a worse outcome. Exploratory endpoint; comparison of baseline score to other points throughout the study.
Time Frame: Up to 52 weeks or early termination
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From first dose through 30 days after last dose of study drug (Up to approximately Week 56)
Description: Safety Sample comprised of participants who received at least one dose of IMP. As prespecified in the SAP, data was analyzed based on the treatments (centanafadine SR 200mg, 400 mg or placebo) received by the participants in the parent double-blind phase 3 trials (405-201-00013 or 405-201-00014), and the centanafadine SR 400 mg received by de novo participants during this current study. Data from 2 parent studies was analyzed and reported in a combined way for rollover participants.
Groups:
- Prior Centanafadine SR 200 mg: Participants who received centanafadine SR 200 mg in the parent double-blind phase 3 studies 405-201-00013 [NCT03605680] or 405-201-00014 [NCT03605836], received centanafadine SR 400 mg TDD in current study, following a dose-escalation schedule. In the current study, participants received centanafadine SR tablets, orally, BID at a starting dose of 200 mg TDD on Day 1 through Day 7, followed by dose-escalation to 400 mg TDD from Day 8 up to Week 52.
- De Novo Centanafadine SR 400 mg: Participants who did not participate in the parents double-blind phase 3 studies 405-201-00013 [NCT03605680] or 405-201-00014 [NCT03605836], and who were eligible for this study received centanafadine SR 400 mg TDD in current study, following a dose-escalation schedule. In the current study, participants received centanafadine SR tablets, orally, BID at a starting dose of 200 mg TDD on Day 1 through Day 7, followed by dose-escalation to 400 mg TDD from Day 8 up to Week 52.
Arm/Group | Prior Centanafadine SR 200 mg | Prior Centanafadine SR 400 mg | Prior Placebo | De Novo Centanafadine SR 400 mg
All-Cause Mortality (participants affected / at risk) | 0/154 | 0/149 | 0/184 | 0/166
Serious Adverse Events (participants affected / at risk) | 1/154 | 1/149 | 7/184 | 3/166
Other Adverse Events (participants affected / at risk) | 59/154 | 49/149 | 81/184 | 61/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prior Centanafadine SR 200 mg (N=154) | Prior Centanafadine SR 400 mg (N=149) | Prior Placebo (N=184) | De Novo Centanafadine SR 400 mg (N=166)
Angina Pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Vertigo Positional (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant Melanoma In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Intentional Self-Injury (Psychiatric disorders) | 0 | 0 | 1 | 1
Mood Swings (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Stress Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prior Centanafadine SR 200 mg (N=154) | Prior Centanafadine SR 400 mg (N=149) | Prior Placebo (N=184) | De Novo Centanafadine SR 400 mg (N=166)
Diarrhoea (Gastrointestinal disorders) | 11 | 6 | 13 | 16
Dry Mouth (Gastrointestinal disorders) | 7 | 6 | 12 | 3
Nausea (Gastrointestinal disorders) | 11 | 7 | 19 | 13
Fatigue (General disorders) | 7 | 4 | 6 | 9
Nasopharyngitis (Infections and infestations) | 8 | 5 | 16 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 7 | 11 | 5
Decreased Appetite (Metabolism and nutrition disorders) | 6 | 7 | 16 | 14
Headache (Nervous system disorders) | 7 | 11 | 14 | 14
Anxiety (Psychiatric disorders) | 8 | 6 | 12 | 11
Insomnia (Psychiatric disorders) | 9 | 10 | 19 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.

DOCUMENTS (2):
  • Study Protocol (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/49/NCT03605849/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT03605849/SAP_001.pdf